CLINICAL TRIAL: NCT02589808
Title: Preoperative Pocket Echocardiography Trial
Acronym: POPPET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15/YH/0333
Record Dates: First submitted 2015-09-29; First posted 2015-10-28 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-09

CONDITIONS: Preoperative Period; Echocardiography
Keywords: pre-operative; transthoracic echocardiography; handheld

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full TTE (Experimental): Full echocardiogram.
  Interventions: Device: Full TTE
- VScan (Experimental): Handheld echocardiogram.
  Interventions: Device: GE Vscan

INTERVENTIONS:
Device: Full TTE — Full transthoracic echocardiogram, with Doppler.
  Arms: Full TTE
Device: GE Vscan — Handheld echo.
  Arms: VScan

SUMMARY:
This study will compare findings using a handheld ultrasound device (GE VScan) with those using a diagnostic ultrasound machine in adult patients referred for transthoracic echo (TTE), prior to non-cardiac surgery at Hammersmith Hospital, London.

The handheld TTE (VTTE) will follow the standard Hammersmith Hospital diagnostic TTE (DTTE) protocol (with the exception of spectral Doppler) and will be reported on a simple 'tick box' form. A different echocardiographer will then perform and report the DTTE as per routine practice. The results from VTTE and DTTE will be directly compared. The echocardiographers performing the VTTE and DTTE are all fully accredited in diagnostic TTE and will be blinded to each others findings.

The study aims to recruit a total of 96 patients with an anticipated study completion date of November 2015.

DETAILED DESCRIPTION:
Handheld echocardiography has become a practical reality with the development of small and highly portable devices. The GE VScan is one such device and a number of studies have examined its diagnostic capabilities in different clinical settings however, no study has examined its capability for screening non-cardiac surgical patients in the preoperative setting. If VTTE could be shown to safely screen patients preoperatively then there is potential to save time and money. DTTE is more costly than VTTE and there are often delays in performing DTTE prior to surgery.

Adult patients > 17 years old who are referred for a preoperative TTE prior to non-cardiac surgery (elective or emergency procedures) are eligible for recruitment. Once an eligible patient is identified verbal and written consent to participate will be obtained.

VTTE will be performed by one of six accredited echocardiographers working in Hammersmith Hospital Echocardiography Department. Based on pilot data and previously published studies it is estimated the VTTE will take between 3 and 7 minutes. The VTTE is reported on a 'tick box' form with the findings separated into significant pathology (red zone) and insignificant pathology or normal findings (black zone).

DTTE will then be performed by a different echocardiographer and a written report prepared as per normal practice. The written DTTE report will be converted to a 'tick box' report enabling direct comparison of VTTE and DTTE.

The primary aim is to assess the ability of the VTTE to detect significant pathology identified on DTTE.

A proportion of DTTE and VTTE will be re-rated to obtain a measure of inter- and intra- observer variability.

ELIGIBILITY:
Inclusion Criteria:

• Adult surgical (non-cardiac) patients referred preoperatively for resting transthoracic echocardiogram

Exclusion Criteria:

• No consent or withdrawal of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petros Nihoyannopoulos, Professor, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, London, East Acton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participant: All Participant went through on full transthoracic echocardiography then GeVscan
Period: Overall Study
Arm/Group | All Participant
Started | 76
Completed | 76
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Echocardiography: Cardiac ultrasound scan.
  Echocardiography: Pocket ultrasound device.
Arm/Group | Echocardiography
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Same Results With GE VScan and Full Transthoracic Echocardiogram
Description: Number of participants who had the same results with both diagnostic device (GE VScan and full transthoracic echocardiogram)
Time Frame: 30min
Measure: Count of Participants; unit: Participants
Groups:
- Echocardiograph: Fully accredited echocardiography laboratory
Arm/Group | Echocardiograph
Number analyzed (Participants) | 76
Participants | 66
Statistical Analysis 1: Comparison: Echocardiograph; Test type: Other; p = 0.0005, Kappa

ADVERSE EVENTS:
Time Frame: 30 min
Arm/Group | Echocardiography
All-Cause Mortality (participants affected / at risk) | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76
Other Adverse Events (participants affected / at risk) | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes